# Designing a Culturally Appropriate Group Navigation Model to Improve Mental and Emotional Health Equity for Spanish-Speaking Latina Women

NCT number: NCT03901430 Unique Protocol ID: 18-305

U54 MD004811 Date: 06-28-2018

### **Principal Investigator**

Julia Meredith Hess, Ph.D., Prevention Research Center, UNM

#### **Research Team:**

Principal Community Mentor and Co-Investigator

Guadalupe Fuentes, Centro Savila

Community Mentor 1

Jacqueline Perez, LCSW, Centro Savila/The Hopkins Center

Community Mentor 2

Alma Olivas, Centro Savila

Research Mentor

Janet Page-Reeves, Ph.D., Family and Community Medicine, UNM

Biostatistician

Cristina Murray-Krezan, MS, CTSC/Internal Medicine, UNM

Community Partner Agency

Centro Savila

Bill Wagner, Ph.D., MSW, Director

Research Assistant

Annette Carrion, UNM Student

Designing a Culturally Appropriate Group Navigation Model to Improve Mental and Emotional Health Equity for Spanish-Speaking Latina Women

#### **Informed Consent for Participation**

06/28/2018

Dr. Julia Hess and health promoter Guadalupe Fuentes and their colleagues from the University of New Mexico and Centro Sávila are conducting a research study with the purpose of investigating how Latina women can improve their mental and emotional health and if a support group and access to community resources can improve the health of participants.

You are being asked to take part in this study because you are a Spanish-speaking Latina woman aged 18 years or older.

Your participation will include being part of a class (which is in the format of a discussion or support group and individual follow-up meetings with the class facilitator, Ms. Fuentes). The time of your involvement will be 6 months. Each class will have about 10 women. There will be three different classes with a total of 30 women. Each class will have 6 sessions. The first 4 sessions will take place once a week (2 hours for each class), followed by a 5<sup>th</sup> class to discuss the results of the class, and then 3 months of individual meetings with the facilitator of the class, Guadalupe Fuentes. After the case management portion is over participants will meet once more for a 6<sup>th</sup> class to discuss the outcomes of the class.

By participating in the class you will also be a member of a study. In order to carry out the study, a member of the study will audio record the class and take notes of the opinions and experiences of the participants. In the analysis of this information we will remove names and identifying information for participants, also ensuring that the recording will be kept in a password protected computer. Only Dr. Julia Hess and members of the study team will have access. One year after the conclusion of the study, the recording will be destroyed.

As part of the study, you will also be asked to complete a survey on your well-being, depression, emotional support, social isolation and empowerment, at two time points: at the beginning of the first and during the last class. Each survey will take between 20 and 30 minutes. Your participation is voluntary and you have the right to decide not to participate. You can decline to respond to any question and withdraw from the study at any time. You will receive a gift card with the value of \$25 to compensate for your time filling out each of the two surveys.

The class is not part of a clinical intervention, and it will not be a part of your medical record. Whether or not you participate in this class will not affect your eligibility access to medical or other resources in the community.

The risks associated with this study are minimal. But some individuals may experience discomfort or loss of privacy when answering questions. Depending on the way you answer some of the questions, we may refer you for mental health services. We can also refer you to mental health resources if you would like to speak to a professional about your condition or if something urgent comes up during the project we will assist you in connecting with appropriate mental health resources. Also, the topics in the class can feel sensitive to some people. We will ask participants to keep within the group any personal information, but we cannot guarantee that everyone will maintain confidentiality. We will do the best we can to ensure that we protect your privacy.

To help us further protect the confidentiality of your data, Dr. Hess has obtained a Certificate of Confidentiality from the National Institutes of Health (NIH). With this certificate, the researchers cannot be forced (for example by court subpoena) to disclose research information that may identify you in any Federal, State, or local civil, criminal, administrative, legislative, or other proceedings. Disclosure will be necessary, however upon request of DHHS or other federal agencies for audit or program evaluation purposes. You should understand that a Certificate of

Confidentiality does not prevent you or a family member from voluntarily releasing information about yourself or your involvement in this research.

The benefit that you may receive from participating in the study is support through the class discussion. The results of the investigation will help us to understand how Latina women can improve their emotional and mental Health. We will publish this information in summary form. If you have any questions about this research project, please feel free to call Dr. Julia Hess at (505) 272-4462. If you have questions regarding your rights as a research subject, you may call the HSC Human Protections Research Office at 505-272-1129.

If you would like to participate in the discussion, please sign below. By signing this form you are agreeing to be part of this study. We will give you a copy of this form.

| | | / |
|---|---|---|
| Name of participant (printed) | Signature of Participant/DATE | |
| <del></del> | | |
| Name of the person witnessing the consent (PRINTED) | Signature of Witness/Date | |

# Diseñando un modelo de navegación grupal culturalmente apropiado para mejorar la equidad en salud mental y emocional para mujeres latinas

#### Abriendo Mis Alas

### Consentimiento Informado para Participación 06/28/2018

La Dra. Julia Hess y la Promotora de Salud y Maestra Guadalupe Fuentes con sus colegas en la Universidad de New México y Centro Sávila están dirigiendo un estudio de investigación, con propósito de investigar como las mujeres Latinas pueden mejorar la salud mental y emocional y si un grupo de apoyo y acceso a los recursos en la comunidad pueden además ayudar a mejorar la salud de las participantes.

Usted está invitada a tomar parte en este estudio porque es una mujer Latina que hable Español y tiene 18 años o más.

Su participación incluye ser parte de una clase (que es en el forma de un grupo de discusión o grupo de apoyo y reuniones individuales con la facilitadora de la clase, Señora Fuentes). El periodo de su involucración seria 6 meses. Cada clase tendrá aproximadamente 10 mujeres. Habrá tres clases diferentes con un total de 30 mujeres. Cada clase tendrá 6 sesiones. Las primeras 4 sesiones se llevaran a cabo una vez a la semana (2 horas para cada clase), seguidas por una 5ª clase para analizar los resultados de la clase, y luego 3 meses de reuniones individuales con el facilitador de la clase, Guadalupe Fuentes.

En participando en la clase, usted tomara parte en un estudio de investigación. Para llevar a cabo el estudio, un miembro del estudio grabará la clase y tomará nota de las opiniones y experiencias de los participantes. Al analizar esta información, retiraremos nombres e información que pueda identificar al participante, asegurando que la grabación se mantenga en una computadora protegida por contraseña: que solo la Dra. Julia Hess y los miembros de su equipo tendrán acceso. Un año después de que concluya la investigación, la grabación será destruida.

También, como parte del estudio, se le pedirá que complete una encuesta sobre su bienestar, la depresión, el apoyo emocional, el aislamiento, y el empoderamiento dos veces, al principio y al final de la clase. Cada encuesta tomara entre 20 y 30 minutos. Su participación en el estudio es voluntaria, y usted tiene el derecho de decidir no participar. Usted puede negarse a responder cualquier pregunta y retirarse del estudio en cualquier momento. Usted recibirá compensación en la forma de una tarjeta de Visa de \$25 por el tiempo que usted ha tomado para cada encuesta. No habrá nombres o información que pueda identificarla con sus respuestas.

Los riesgos asociados con ésta investigación son mínimos. Algunas personas pueden sentirse incomodas o temerosas de la posible perdida de privacidad al contestar nuestras preguntas en las encuestas. Dependiendo de la forma en que responda algunas de las preguntas, podemos referirlo a servicios de salud mental. Además podremos brindarle información sobre los recursos de salud mental, por si usted quiere hablar con algún profesional acerca de su condición o si surge algo durante la clase que le gustaría abordar con un profesional de la salud mental afuera de la clase.

También, de lo que se hable en el grupo de apoyo, algunas personas podrían ser consideradas sensitivas. Pediremos a los participantes mantener la confidencial sobre cualquier información personal dentro del grupo, pero no podemos garantizarlo fuera de el. Nosotros haremos lo mejor que podamos para asegurarnos que su información se mantenga en privado.

Para ayudarnos a proteger la confidencialidad de sus datos, la Dra. Julia Hess ha obtenido un Certificado de Confidencialidad del Instituto Nacional de Salud (National Institute of Health – NIH). Con este certificado los investigadores no pueden ser forzados (por ejemplo por una citación judicial) a revelar información sobre la investigación que pueda identificarlo en cualquier corte Federal, Estatal, local o civil, criminal, administrativa, legislativa, o cualquier otro procedimiento. El revelar información solo será necesario a la petición del DHHS o alguna otra agencia federal, cual propósito sea auditivo o sobre algún programa de evaluación. Usted debe de entender que el Certificado de Confidencialidad no preventa que usted o algún miembro de su familia comparta información sobre usted o sobre su participación en esta investigación voluntariamente.

El beneficio es que usted puede recibirá del estudio es el apoyo a través del grupo de discusión. Los resultados de la investigación nos ayudarán a entender cómo las mujeres latinas pueden mejorar su salud emocional y mental. Estos se publicarán en forma resumida.

Si usted tiene alguna pregunta sobre esta investigación, por favor de contactar a la Dra. Julia Hess al (505) 272-4462 o si tiene alguna pregunta sobre sus derechos como un participante de investigación. Si usted quisiera hablar con alguien más aparte del grupo de investigación, por favor llame a la Oficina de Protección de Investigación en Humanos al número 505-272-1129.

Si usted quiere participar en este grupo de discusión, por favor firme abajo. Al firmar este formulario usted está aceptando ser parte de este estudio. Le daremos una copia de este formulario.

| Nombre del Participante (en letra de molde) | Firma del Participante/ | / |
|---|---|---|
| Nombre de la Persona que explica el formulario de consentimiento | Firma de la Persona | /_<br>Fecha |